CLINICAL TRIAL: NCT03392597
Title: Testing the Efficacy of a Strengths-Based Curriculum to Reduce Risk for Future Sexual Violence Perpetration Among Middle School Boys
Brief Title: Preventing Sexual Violence Among Middle School Boys With a Strengths-Based Curriculum
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: New York State Department of Health (Other Government)
Collaborators: Cornell University (Other)
Responsible Party: Principal Investigator, Janis Whitlock, Research Scientist, Cornell University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CE002834
Record Dates: First submitted 2017-08-03; First posted 2018-01-08 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Sexual Violence

STUDY DESIGN:
Intervention Model Description: Waitlist control design in which matched sites are randomly assigned to an intervention or waitlist control group to implement and evaluate the Brothers as Allies program. Intervention groups will participate in the Brothers as Allies program from the Council for Boys and Young Men. Waitlist control groups will participate in programming-as-usual until implementation with the intervention groups is complete, at which point they will receive the intervention. All participants will complete surveys at baseline, immediate post-intervention, and at 3 and 6 months post-intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brothers as Allie (Experimental): Brothers as Allies is a strengths-based group approach to promote boys' and young men's safe and healthy passage through the pre-teen and adolescent years by addressing rigid beliefs and norms about masculinity that are harmful to the health, safety, relationships and opportunities of boys and young men. Groups of six to ten boys of similar age and development meet weekly with one or two facilitators for 1.5 to 2 hours for ten or more weeks. Meetings include warm up activities, an opportunity for check-in, experiential activities that address gender relevant topics (e.g., group challenges, games, skits, role plays), and a reflection and group dialogue component.
  Interventions: Behavioral: Brothers as Allies
- Programming-as-Usual (Active Comparator): Usual programming implemented in afterschool programs.
  Interventions: Behavioral: Programming-as-Usual

INTERVENTIONS:
Behavioral: Brothers as Allies — Strengths-based group approach to promote boys' and young men's safe and healthy passage through the pre-teen and adolescent years.
  Arms: Brothers as Allie
Behavioral: Programming-as-Usual — Usual afterschool programming.
  Arms: Programming-as-Usual

SUMMARY:
This research will examine if participation in a strengths-based curriculum, the Brothers as Allies program adapted from the Council for Boys and Young Men, reduces risk for future sexual violence perpetration among middle school-aged boys in New York State.

DETAILED DESCRIPTION:
Using a longitudinal waitlist control design, this study will evaluate the efficacy of a strengths-based curriculum, the Brothers as Allies program from the Council for Boys and Young Men, to reduce risk for future sexual violence perpetration with middle school-aged boys (ages 12-14) in New York State. This research will examine if participation in the program decreases negative behaviors (such as later sexual violence perpetration and sexual aggression) and increases positive behaviors (such as bystander intervention and caring/cooperative behaviors) amongst program participants, in comparison to participants who participate in programming-as-usual. Other potential moderators and outcomes linked to sexual violence victimization and sexual assault perpetration (including attitudes related to gender roles, acceptance of sexual violence, and interpersonal relationships) will also be measured. The research team will also assess the extent to which the curriculum, when implemented with fidelity and quality, leads to improved relationships and stronger connections with adults in afterschool or other community-based youth-program settings. All participants will complete surveys at baseline, immediate post-intervention, and at 3 and 6 months post-intervention. Finally, the investigators will also assess the implementation factors which impact the efficacy of this program, such as fidelity and quality of program delivery. The research team hypothesizes participants in the Brothers as Allies program will show post-intervention decreased sexual violence perpetration, less acceptance of sexual violence, less stereotypic gender role attitudes, greater youth-adult connectedness, and increased bystander intervention, caring, and cooperation behaviors compared to peers in the non-intervention group. In order to complete this work, the research team is collaborating with the New York Rape Prevention and Education (RPE)-funded Regional Centers for Sexual Violence Prevention and a Research Advisory Board of community members and professionals from New York State.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be males of middle school age (12-14 years), participating in afterschool/youth programming at one of the intervention or control sites.

Exclusion Criteria:

* None.

Ages: 12 Years to 14 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Middle school-aged boys
Enrollment: 720 (Estimated)
Dates: Start 2017-07-26 (Actual); Primary Completion 2020-07-24 (Estimated); Study Completion 2020-09-29 (Estimated)

PRIMARY OUTCOMES:
Sexual violence perpetration (Koss et al., 2006) | 3 months
  This will be measured by items from a widely used measure of sexual violence perpetration behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Janis Whitlock, PhD, Principal Investigator — Cornell University
Locations (1):
- Planned Parenthood of Central and Western New York, Rochester, New York, United States